CLINICAL TRIAL: NCT04528407
Title: Follow-up Study for Patients Having Received FluBHPVE6E7 in Clinical Studies
Brief Title: BS-FU01 Follow-Up Study of FluBHPVE6E7 Study Subjects
Status: Completed | Type: Observational
Sponsor: BlueSky Immunotherapies GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: BS-FU01
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Safety Issues; HPV Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Observation; Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for determination of the immune response Nasal secretion and blood samples for biodistribution Cervical smear for cytology and HPV test Urine for Pregnancy test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation without intervention — This study is a follow-up study without intervention.

SUMMARY:
This is a follow-up study for patients treated with FluBHPVE6E7 in previous interventional studies.

DETAILED DESCRIPTION:
BS-FU01 is a follow-up study for patients treated with FluBHPVE6E7 in previous phase 1 and 2 interventional studies. The aim of the follow-up study is to assess the safety and immunogenicity of FluBHPVE6E7, changes in the HPV infection status, cervical cytology, and biodistribution after treatment with FluBHPVE6E7 in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient who enrolled in previous phase 1 or 2 clinical studies of FluBHPVE6E7
* Negative pregnancy test at baseline
* Written informed consent

Exclusion Criteria:

* Pregnancy, breastfeeding

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who enrolled in previous phase 1 or 2 clinical studies of FluBHPVE6E7
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (type, frequency, severity). | 1 year
  To assess the safety and tolerability of FluBHPVE6E7 by monitoring the type, frequency, and severity of AEs

SECONDARY OUTCOMES:
Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) following FluBHPVE6E7 administration | 1 year
  To evaluate of the induction of systemic vector-specific antibodies by HAI assay
Induction of HPV-specific T-cell response following FluBHPVE6E7 administration | 1 year
  To evaluate the induction of HPV16 E6- and E7-specific T-cells (percent %) by IFN-gamma ELISPOT analysis
Induction of HPV-specific CD4+ and CD8+ T-cells following FluBHPVE6E7 administration | 1 year
  To evaluate the induction of HPV16 E6- and E7 specific T-cells (percent %) by ICS and FACS analysis
Local HPV clearance | 1 year
  To evaluate the status of HPV-16 infection by HPV test (yes or no)
Cervical cytology | 1 year
  To evaluate changes in cervical cytology by Pap smear. Results are reported as Pap results according to the Bethesda System
Biodistribution: Detection of FluBHPVE6E7 in blood samples | 1 year
  To evaluate the presence of FluBHPVE6E7 by quantification of FluBHPVE6E7 genome copies in blood samples by RT-qPCR (copies per ml blood)
Biodistribution: Detection of FluBHPVE6E7 in nasal secretions | 1 year
  To evaluate the presence of FluBHPVE6E7 by qualitative real-time PCR assay specific for influenza B virus (positive or negative)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided